CLINICAL TRIAL: NCT00952640
Title: Making Maternal Post-partum Vitamin A Supplementation Effective: The Role of Timing and Inflammation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Thrasher Research Fund (Other); University of Copenhagen (Other); National Institute of Nutrition, Vietnam (Other Government)
Responsible Party: Principal Investigator, Frank Wieringa, Senior Rechercher, Institut de Recherche pour le Developpement
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: VitA_PP
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Healthy Women Giving Birth to Singleton Infants
Keywords: vitamin A; post-partum; infant; acute phase response
MeSH Terms: conditions — Acute-Phase Reaction | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin A directly post-partum (Active Comparator): 200.000 IU of vitamin A within 3 days of delivery
  Interventions: Dietary Supplement: vitamin A
- vitamin A delayed (Experimental): 200.000 IU vitamin A 6 weeks post-partum
  Interventions: Dietary Supplement: vitamin A

INTERVENTIONS:
Dietary Supplement: vitamin A — high dose vitamin A, 200.000 IU

SUMMARY:
Background:

Vitamin A is of utmost importance for health and survival of children. A recent series in The Lancet on maternal and child health put vitamin A deficiency at the top of most important micronutrient deficiencies, responsible for more than 600.000 child deaths/year worldwide. Vitamin A status of mothers and infants is closely linked. Hence, a mother with vitamin A deficiency cannot give enough vitamin A to her fetus to build stores during the last months of pregnancy, and will also have insufficient amounts of vitamin A in her breast milk, resulting in a high risk for vitamin A deficiency in her newborn infant. The World Health Organization (WHO) has implemented several strategies to fight vitamin A deficiency in mothers and children. One of these is to give women after delivery a high dose vitamin A supplement, to improve vitamin A status of mother and, via breast milk, her infant. Surprisingly however, several recent studies investigating the effect of a high dose vitamin A supplement for mothers directly after birth found no effect on vitamin A status in infants 6 months of age. In contrast, earlier studies in Bangladesh and Indonesia, in which women received a high dose vitamin A supplement somewhere in the first 6 weeks after delivery, reported a large impact on vitamin A status in the infants at 6 mo of age. The WHO recommendation on post-partum vitamin A supplementation was based on these earlier studies from Bangladesh and Indonesia. The more recent studies suggest however that this intervention is not effective, and that millions of women currently receive a high dose vitamin A supplement without clear benefits for vitamin A status in either the women or their children.

The human body reacts to infection or injury with an inflammatory response, which kicks off with the acute phase response. The acute phase response helps the body to fight the infection. It is characterized by many altered physiological processes, including changed availability of vitamins and minerals. Recently, we found that delivery in itself causes a major acute phase response. We have formed the hypothesis that the acute phase response initiated by delivery prevents the high dose vitamin A supplement given to the mother directly after delivery from being absorbed and from being available for breast milk. If this is true, the current WHO recommendation to give the vitamin A within the first 6 weeks post-partum should be changed to giving the vitamin A 4 - 6 weeks post-partum instead, to allow the acute phase response induced by delivery to fade.

Objective(s) and Hypothesis(es):

The main objective is to improve the effectiveness of the current WHO policy of vitamin A supplementation after delivery to improve vitamin A status and health of mothers and their infants.

Methodology:

In a randomized, placebo-controlled, double-blind trial, 400 women will receive a high dose of vitamin A (200.000 IU) within 6 weeks of delivery, as recommended by WHO. Half of the women will receive the vitamin A directly after delivery (within 3 days, current practice), whereas the other women will receive the vitamin A 6 weeks after delivery. To guarantee blinding, women will receive a placebo capsule if they are not receiving a vitamin A capsule.

Main outcomes will be maternal and infant vitamin A status 6 months post-partum and the time-course of the acute phase response, to establish the optimal time after delivery for the initiation of the vitamin A supplementation.

Secondary outcomes will be the morbidity of the infants during the first 6 months of life and growth performance of the infants at 6 mo of age.

Potential Impact:

The results of this study will enable WHO to improve the effectiveness of the current WHO recommendations concerning post-partum vitamin A supplementation. If our hypothesis is true, postponing the timing of the post-partum vitamin A supplement from directly after delivery to 6 week post-partum, will significantly increased the availability of the supplement for the mother. This will increase the vitamin A status of both mother and infant. Moreover, there are several significant implications for global health policies, with important consequences for infant survival worldwide by reducing morbidity and mortality from infectious diseases during the first 6 months of life. Results of the study will also have important consequences for other micronutrient health programs, such as vitamin A supplementation for children above 6 months of age and iron supplementation in areas with endemic malaria, as these are also subject to the effects of the acute phase response

DETAILED DESCRIPTION:
Background. Undernutrition causes over 3.5 million child deaths a year, with vitamin A deficiency alone responsible for almost 0.6 million child deaths per year1. Vitamin A supplementation of children above 6 months of age has been shown to reduce overall mortality by 23%. The effect of vitamin A supplementation in newborns on morbidity and mortality is less clear, with three studies in India, Indonesia and Nepal showing reductions in neonatal mortality of 22%, 64% and 15% respectively, but with 2 other trials in Africa reporting no effect. In view of the expected health benefits of improved vitamin A status of infants, WHO currently recommends that women should receive a high dose (200.000 IU ) of vitamin A within the first 6 weeks postpartum, in order to improve maternal vitamin A status, the vitamin A content of breast milk, and thereby the vitamin A status of their infants. However, several recent trials in which women received 200.000 IU vitamin A directly post-partum, reported no improvement in vitamin A status of either mother or her infant at 6 mo of age, not even after doubling the dose to 400.000 IU. In these studies vitamin A was given within a week of delivery, the current typical practice even though WHO actually states a window of 6 weeks after delivery. In contrast, 2 earlier studies in Bangladesh and Indonesia reported a large impact of post-partum maternal supplementation on vitamin A status in infants at 6 mo of age. In these studies, women received a high dose vitamin A supplement not directly post-partum, but somewhere in the first 6 weeks after delivery. The WHO recommendation on maternal post-partum vitamin A supplementation was based on the effects observed in these earlier studies, but the more recent studies suggest now that this intervention is not effective, and that millions of women are receiving a high dose vitamin A supplement without clear benefits for vitamin A status of either the women or their children. The difference in timing between the earlier studies and the recent studies of giving the vitamin A may hold the key, and we believe we have identified the biological reason why timing of the supplementation could be of the utmost importance: the inflammatory response to delivery.

Delivery induces a considerable physiological inflammatory response, with a distinct acute phase response, of the same magnitude as seen for instance in pulmonary tuberculosis patients. We believe that the lack of effect of the current practice of giving a high dose vitamin A supplement directly post-partum is due to the acute phase response induced by the delivery, and that the intervention would be successful if the supplementation was given after the acute phase response has faded away after 3 - 6 weeks. There is currently no data available on the vitamin A bioavailability in lactating women, but a study in Zambian pre-school children investigated the effectiveness of a high dose vitamin A supplementation campaign in children, and showed that this was only successful in children without inflammation. Children who had signs of inflammation had no increase in vitamin A status. Inflammation and the accompanying acute phase response are also known to affect the availability of other micronutrients besides vitamin A, such as iron and zinc.

Objective(s) and Hypothesis(es):

Hypothesis The acute phase response (APR) induced by delivery reduces vitamin A bioavailability, and interferes with current maternal post-partum high dose vitamin A supplementation programs worldwide.

Objective 1 To determine the effects of the acute phase response on vitamin A bioavailability.

Objective 2 To determine the time course of the acute phase response after delivery.

Overall goal To improve the effectiveness of the current WHO recommendation of post-partum maternal high dose vitamin A supplementation by determining the optimal timing for supplementation in relation to the post-partum APR.

Design and Methods:

A randomised, placebo-controlled, double-blind trial in 400 women, comparing the effects of the recommended dose of 200.000 IU of vitamin A given within the first week post-partum (current practice, 200 women) with the effect when given at 6 weeks post-partum, which is still within the WHO recommended intervention window (200 women). Main outcomes will be maternal and infant vitamin A status 6 months post-partum, breast milk vitamin A concentrations and the time-course of acute phase response, to establish the optimal time after delivery for vitamin A supplementation. Secondary outcomes will be morbidity of the infants during the first 6 months of life and anthropometrical indices of the infants at 6 mo of age.

Potential Impact:

If our hypothesis is true, the current global health strategy of postpartum vitamin A supplementation to improve vitamin A status of mothers and infants can be made effective just by changing the timing. This will have significant implications for global health policies, with important consequences for infant survival worldwide by improving vitamin A status and reducing morbidity and mortality from infectious diseases during the first 6 months of life. Moreover, results of the study will have important consequences for other micronutrient health programs, such as vitamin A supplementation for children above 6 months of age and iron or zinc supplementation programs, as these are also affected by the acute phase response. Overall, the results of this research will contribute to improving child survival worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women giving birth to a singleton infant.

Exclusion Criteria:

* Women giving birth to infants weighing < 1500 gram (very low birth weight infant) will be excluded.
* Also excluded will be twin pregnancy, because of different growth patterns of the infants and congenital abnormalities interfering with normal growth.
* Furthermore, women indicating that they are planning not to breast feed their baby will be excluded, as well as women who experience delivery complications which result in prolonged (> 3 days) hospital stay.
* Complications such as eclampsia or excessive blood loss will be registered, but will not be a reason for exclusion per se.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
vitamin A status of lactating women 6 mo post-partum vitamin A status of infants 6 mo of age acute phase proteins concentrations (CRP, AGP) at several time-points during the first 6 mo post-partum | several times points during the first 6 mo post-partum (different time points for different indicators)
plasma retinol 6 mo post-partum (women and infants), breast milk retinol (6 weeks, 4 mo and 6 mo post-partum), liver retinol stores of infants 6 mo post-partum acute phase proteins, at 2 weeks, 6 weeks, 4 mo and 6 mo post-partum (women) | 2 and 6 weeks, 4 mo and 6 mo post-partum

SECONDARY OUTCOMES:
morbidity infants during the first 6 mo of life anthropometry at 6 mo post-partum | 6 mo of age

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Nutrition, Hanoi, Vietnam

REFERENCES:
- [Background] Friis H, Range N, Braendgaard Kristensen C, Kaestel P, Changalucha J, Malenganisho W, Krarup H, Magnussen P, Bengaard Andersen A. Acute- phase response and iron status markers among pulmonary tuberculosis patients: a cross-sectional study in Mwanza, Tanzania. Br J Nutr. 2009 Jul;102(2):310-7. doi: 10.1017/S0007114508162122. Epub 2009 Jan 28. PMID 19175946
- [Background] Ayah RA, Mwaniki DL, Magnussen P, Tedstone AE, Marshall T, Alusala D, Luoba A, Kaestel P, Michaelsen KF, Friis H. The effects of maternal and infant vitamin A supplementation on vitamin A status: a randomised trial in Kenya. Br J Nutr. 2007 Aug;98(2):422-30. doi: 10.1017/S0007114507705019. Epub 2007 Mar 29. PMID 17391562
- [Background] Wieringa FT, Dijkhuizen MA, van der Meer JW. Maternal micronutrient supplementation and child survival. Lancet. 2008 May 24;371(9626):1751-2. doi: 10.1016/S0140-6736(08)60758-8. No abstract available. PMID 18502294
- [Background] Dijkhuizen MA, Wieringa FT, West CE, Muhilal. Zinc plus beta-carotene supplementation of pregnant women is superior to beta-carotene supplementation alone in improving vitamin A status in both mothers and infants. Am J Clin Nutr. 2004 Nov;80(5):1299-307. doi: 10.1093/ajcn/80.5.1299. PMID 15531679